CLINICAL TRIAL: NCT04737980
Title: Liposomal Bupivacaine Plus Bupivacaine Peripheral Nerve Blockade Versus Ropivacaine Plus Dexamethasone Peripheral Nerve Blockade for Arthroscopic Rotator Cuff Repair: a Prospective Randomized Trial
Brief Title: Liposomal Bupivacaine Plus Bupivacaine Peripheral Nerve Blockade Versus Ropivacaine Plus Dexamethasone Peripheral Nerve Blockade for Arthroscopic Rotator Cuff Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery Florida (Other)
Responsible Party: Principal Investigator, ryan simovitch, Director-Shoulder Service, Hospital for Special Surgery Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JMC0023RSOP
Record Dates: First submitted 2021-01-23; First posted 2021-02-04 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Rotator Cuff Tears; Shoulder Pain
Keywords: peripheral nerve block; interscalene nerve block; bupivacaine; liposomal bupivacaine; ropivacaine; dexamethasone
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain | interventions — Bupivacaine; Ropivacaine; Dexamethasone

STUDY DESIGN:
Intervention Model Description: This study utilized two parallel arms for intervention. Participants were randomized to ultrasound guided PNB with liposomal bupivacaine combined with bupivacaine or PNB with ropivacaine combined with dexamethasone.
Who Masked: Outcomes Assessor
Masking Description: The participant was informed of which arm they were in after random draw as this information may have been important in the event they experienced side effects and needed to guide physician care at outside facilities. The anesthesiologist could not be masked regarding arm as the appearance of the medicine injected in both arms of the study was visibly different. The outcome assessor was masked by unique identifiers being applied to participants and outcome data kept separate from intervention arm until final analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental Group: Interscalene block with liposomal bupivacaine combined with bupivacaine (Experimental): Interscalene nerve block was performed utilizing ultrasound guidance with infiltration of 10 ml of liposomal bupivacaine 1.3% (133 mg) combined with 10 ml of 0.5% bupivacaine hydrochloride.
  Interventions: Drug: Liposomal bupivacaine; Drug: Bupivacaine Hcl 0.5% Inj
- Control Group: Interscalene block with ropivacaine combined with dexamethasone (Active Comparator): Interscalene nerve block was performed utilizing ultrasound guidance with infiltration of 30ml of 0.5% ropivacaine combined with a 2 ml volume of 8mg of dexamethasone.
  Interventions: Drug: Ropivacaine 0.5% Injectable Solution; Drug: Dexamethasone

INTERVENTIONS:
Drug: Liposomal bupivacaine — Injection of 10 ml of liposomal bupivacaine 1.3% (133 mg) for ultrasound guided interscalene block
  Other Names: Exparel
  Arms: Experimental Group: Interscalene block with liposomal bupivacaine combined with bupivacaine
Drug: Bupivacaine Hcl 0.5% Inj — Injection of 10 ml of 0.5% bupivacaine hydrochloride as admixture for ultrasound guided interscalene block
  Arms: Experimental Group: Interscalene block with liposomal bupivacaine combined with bupivacaine
Drug: Ropivacaine 0.5% Injectable Solution — Injection of 30 ml of ropivacaine 0.5% injectable solution for ultrasound guided interscalene block
  Arms: Control Group: Interscalene block with ropivacaine combined with dexamethasone
Drug: Dexamethasone — Injection of 8mg (2ml) dexamethasone injectable as admixture
  Arms: Control Group: Interscalene block with ropivacaine combined with dexamethasone

SUMMARY:
This study is a comparison of analgesia effect from peripheral nerve blockade (PNB) with liposomal bupivacaine combined with bupivacaine compared to PNB with ropivacaine combined with dexamethasone for arthroscopic rotator cuff repair.

DETAILED DESCRIPTION:
Arthroscopic rotator cuff repair(ARCR) addresses dysfunction and pain in individuals with rotator cuff tears who have failed conservative management. These procedures are typically performed in an outpatient setting. Single shot PNB with long acting local anesthetics have become the foundation of modern multimodal analgesia protocols. The reported analgesic benefits of PNB for shoulder surgery include reduced pain scores, opioid consumption, post-operative nausea and vomiting, improved postoperative recovery and improvement of patient satisfaction. However, standard PNB with bupivacaine or ropivacaine have been associated with rebound pain resulting in a sudden onset of pain that can be refractory to treatment and often necessitates the use of significant quantities of opioids.

Side effects of opioid consumption include nausea, vomiting, sedation, constipation, respiratory depression, hypotension, ileus, urinary retention, dehydration and addiction. It is therefore desirable to minimize the requirement for opioid consumption after ARCR.

Liposomal bupivacaine injectable suspension and its potential use for PNB has been a recent topic of interest in an effort to provide patients with longer acting pain control after shoulder surgery compared to the use of bupivacaine or ropivacaine. Liposomal bupivacaine has a delayed onset of action so its practical use for PNB for ARCR requires the additive of bupivacaine to reduce pain during and immediately after surgery as a bridge to the onset of liposomal bupivacaine.

The purpose of this study is to determine if PNB utilizing liposomal bupivacaine combined with bupivacaine performs favorably to standard PNB with ropivacaine combined with dexamethasone. Primary and secondary outcomes will be assessed including worst pain reported postoperatively on a numeric rating scale(NRS), postoperative opioid consumption reported as oral morphine equivalent dosage(OMED) and the overall benefit of anesthesia (OBAS) as reported by the OBAS score.

The hypothesis of this study is that PNB with liposomal bupivacaine combined with bupivacaine will translate to lower postoperative daily NRS pain scores, decreased daily and total OMED consumed and lower OBAS scores compared to PNB with ropivacaine combined with dexamethasone over the first 8 days following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Full thickness tears of the Supraspinatus tendon
* Combined full thickness tears of the Supraspinatus and Infraspinatus tendon

Exclusion Criteria:

* Age < 18
* Revision surgery
* Chronic opioid use (>3 months prior to surgery)
* Allergy to local anesthetics or opioids
* Workers compensation or medical legal claim
* Pulmonary disease
* NSAID intolerance
* Neurologic deficit of operative upper extremity
* Concomitant full thickness subscapularis tear

  * 2 tendon rotator cuff tear

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Daily morphine milligram equivalents of opioid | up to 8 days
  Daily opioid consumption reported as OMED
Total opioid consumption in morphine milligram equivalents | 8 day period
  Total opioid consumption for entire 8 days after surgery
Participant reported "worst pain" level on a numeric rating scale after surgery | up to 8 days
  Worst pain level experienced as reported on a numeric rating scale by a participant for each preceding 24 hour period. 0 on numeric rating scale denoting no pain and 10 denoting worst possible pain.
Overall benefit of anesthesia score (OBAS) | up to 8 days
  Overall benefit of anesthesia score (OBAS) as reported by a participant for each preceding 24 hour period. OBAS is a numeric rating scale. A lower value denotes better pain control and less side effects from anesthesia. Range of scores from 0 to 28.

SECONDARY OUTCOMES:
Change in pain from baseline | up to 8 days
  Participant reported change in "worst pain" level on numeric rating scale from baseline (preoperative) "worst pain" to "worst pain" reported on each day after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- HSS Florida, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Uquillas CA, Capogna BM, Rossy WH, Mahure SA, Rokito AS. Postoperative pain control after arthroscopic rotator cuff repair. J Shoulder Elbow Surg. 2016 Jul;25(7):1204-13. doi: 10.1016/j.jse.2016.01.026. Epub 2016 Apr 11. PMID 27079219
- [Result] Hussain N, Brull R, Sheehy B, Essandoh MK, Stahl DL, Weaver TE, Abdallah FW. Perineural Liposomal Bupivacaine Is Not Superior to Nonliposomal Bupivacaine for Peripheral Nerve Block Analgesia. Anesthesiology. 2021 Feb 1;134(2):147-164. doi: 10.1097/ALN.0000000000003651. PMID 33372953
- [Result] Abdallah FW, Halpern SH, Aoyama K, Brull R. Will the Real Benefits of Single-Shot Interscalene Block Please Stand Up? A Systematic Review and Meta-Analysis. Anesth Analg. 2015 May;120(5):1114-1129. doi: 10.1213/ANE.0000000000000688. PMID 25822923
- [Result] Namdari S, Nicholson T, Abboud J, Lazarus M, Steinberg D, Williams G. Interscalene Block with and without Intraoperative Local Infiltration with Liposomal Bupivacaine in Shoulder Arthroplasty: A Randomized Controlled Trial. J Bone Joint Surg Am. 2018 Aug 15;100(16):1373-1378. doi: 10.2106/JBJS.17.01416. PMID 30106818
- [Result] Namdari S, Nicholson T, Abboud J, Lazarus M, Steinberg D, Williams G. Randomized Controlled Trial of Interscalene Block Compared with Injectable Liposomal Bupivacaine in Shoulder Arthroplasty. J Bone Joint Surg Am. 2017 Apr 5;99(7):550-556. doi: 10.2106/JBJS.16.00296. PMID 28375887
- [Result] Kolade O, Patel K, Ihejirika R, Press D, Friedlander S, Roberts T, Rokito AS, Virk MS. Efficacy of liposomal bupivacaine in shoulder surgery: a systematic review and meta-analysis. J Shoulder Elbow Surg. 2019 Sep;28(9):1824-1834. doi: 10.1016/j.jse.2019.04.054. Epub 2019 Jul 16. PMID 31324503
- [Result] Yan Z, Chen Z, Ma C. Liposomal bupivacaine versus interscalene nerve block for pain control after shoulder arthroplasty: A meta-analysis. Medicine (Baltimore). 2017 Jul;96(27):e7226. doi: 10.1097/MD.0000000000007226. PMID 28682872
- [Result] Patel MA, Gadsden JC, Nedeljkovic SS, Bao X, Zeballos JL, Yu V, Ayad SS, Bendtsen TF. Brachial Plexus Block with Liposomal Bupivacaine for Shoulder Surgery Improves Analgesia and Reduces Opioid Consumption: Results from a Multicenter, Randomized, Double-Blind, Controlled Trial. Pain Med. 2020 Feb 1;21(2):387-400. doi: 10.1093/pm/pnz103. PMID 31150095
- [Result] Wang K, Zhang HX. Liposomal bupivacaine versus interscalene nerve block for pain control after total shoulder arthroplasty: A systematic review and meta-analysis. Int J Surg. 2017 Oct;46:61-70. doi: 10.1016/j.ijsu.2017.08.569. Epub 2017 Aug 24. PMID 28843463